CLINICAL TRIAL: NCT04442945
Title: A Double-blind, Randomized, Placebo-controlled, Phase 1 Safety and Tolerability, and Pharmacokinetics Study of ANAVEX3-71
Brief Title: Phase 1 Study of ANAVEX3-71
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Collaborators: Anavex Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANAVEX3-71-001
Record Dates: First submitted 2020-06-17; First posted 2020-06-23 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANAVEX3-71 Oral (Experimental): Up to four single ascending doses of ANAVEX3-71 administered orally
  Interventions: Drug: ANAVEX3-71
- Placebo arm Oral (Placebo Comparator): Placebo administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ANAVEX3-71 — Active oral dose of ANAVEX3-71
  Arms: ANAVEX3-71 Oral
Drug: Placebo — Oral placebo
  Arms: Placebo arm Oral

SUMMARY:
A first in human phase 1 study in healthy volunteers to assess ANAVEX3-71 safety, tolerability, bioavailability, pharmacokinetics, and pharmacodynamics

DETAILED DESCRIPTION:
This is a first-in-human Phase 1 study designed to investigate the safety, tolerability, PK, PD and bioavailability of orally administered ANAVEX3-71 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female between 18 and 55 years of age, inclusive.
* Body mass index (BMI) between 19-28 kg/m2 and within a body weight of ≥ 60 kg and ≤ 120 kg.
* Female subjects must be of non-childbearing potential (defined as postmenopausal for at least 2 years or surgically sterile at least 6 months prior to dosing) or must be using adequate contraception.
* Subject is judged by the investigator to be in generally good health at screening based upon the results of a medical history, physical examination, laboratory profile, and 12-lead electrocardiogram (ECG).
* Non-smoker (no tobacco use within past 3 months).
* Subject is willing to comply with the study protocol, in the investigator's judgement.

Exclusion Criteria:

* Subject has a history or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, dermatological, neurological, psychiatric, hematological (including myelosuppression and bleeding disorders) or immunological/autoimmune disorder(s), and/or any condition that could constitute a potential safety risk factor or could alter the absorption, distribution, metabolism or elimination of the study drugs.
* Positive test result on Hepatitis B surface antigen (HBsAg) or is Hepatitis C virus antibody (HCV-Ab) positive or positive HIV-1 and/or -2 serology.
* Subject has a history of chronic alcohol abuse within the last 2 years, or has a positive alcohol test or is known to have excessive alcohol intake.
* History of substance abuse, known drug addiction, or positive test for drugs of abuse.
* Subject has participated in another clinical trial of an investigational drug (or a medical device) within the last 3 months or is currently participating in another trial of an investigational drug (or a medical device).
* Female subject who is pregnant or lactating or planning a pregnancy.
* A history of major mental illness that in the opinion of the Investigator may affect the ability of the subject to participate in the study (psychosis is to be disqualified).
* Subject has a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the subject at undue risk.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability of ANAVEX3-71 measured by number of subjects with adverse events and Dose Limiting Adverse Event (DLAEs) Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 30 days
  Incidence of adverse events and dose limiting Adverse Events during the DLAE observation period and/or study treatment periods.
Pharmacokinetics (PK) of ANAVEX3-71 | 30 days
  Serum concentration of ANAVEX3-71 at specified time points
Maximum plasma concentration (Cmax) for ANAVEX3-71 | 30 days
  Evaluate Cmax for serum concentration of ANAVEX3-71 at specified time points
Area under the curve concentration (AUC) for ANAVEX3-71 | 30 days
  Evaluate AUC for serum concentration of ANAVEX3-71 at specified time points

SECONDARY OUTCOMES:
Effect on ECG, including the ECG QT Interval | 30 days
  To characterize the effect on ECG, including the ECG QT Interval for ANAVEX3-71

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: Undecided